CLINICAL TRIAL: NCT00266214
Title: A Randomized, Double-Blind Study Comparing the Safety and Efficacy of the Lidocaine Patch 5% With Placebo in Patients With Pain From Carpal Tunnel Syndrome
Brief Title: Safety and Efficacy of Lidoderm (Lidocaine Patch 5%) in Treating Moderate to Severe Pain Associated With Carpal Tunnel Syndrome
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Endo Clinical Trials Response Center, Endo Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EN3272-301
Record Dates: First submitted 2005-12-15; First posted 2005-12-16 (Estimated); Last update posted 2011-06-14 (Estimated); Status verified 2011-06

CONDITIONS: Carpal Tunnel Syndrome
Keywords: lidocaine patch 5%; Lidoderm; carpal tunnel syndrome; pain; nerve compression injury; topical analgesic
MeSH Terms: conditions — Carpal Tunnel Syndrome; Pain; Neuroma | interventions — Lidoderm

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Lidocaine Patch 5% (Experimental): 1 patch applied topically to the volar aspect of each affected wrist daily, 2-4 hours before bedtime.
  Interventions: Drug: lidocaine patch 5%
- Placebo (Placebo Comparator): 1 patch applied topically to the volar aspect of each affected wrist daily, 2-4 hours before bedtime.
  Interventions: Drug: lidocaine patch 5%

INTERVENTIONS:
Drug: lidocaine patch 5% — 1 patch applied topically to the volar aspect of each affected wrist daily, 2-4 hours before bedtime
  Other Names: Lidoderm

SUMMARY:
The purpose of this study is to evaluate the analgesic efficacy and safety of the lidocaine patch 5% compared to placebo in patients with moderate to severe pain associated with carpal tunnel syndrome.

DETAILED DESCRIPTION:
Patients with carpal tunnel syndrome (CTS)as determined by electrodiagnostic testing and moderate to severe pain will be randomized to receive either the lidocaine patch 5% or placebo patch q24h. The total duration of the double-blind treatment phase of the study will be 8 weeks.

At baseline and at periodic visits to the clinic, patients will perform pain and functionality assessments. Patients with bilateral CTS will identify the "index" wrist (i.e., the more painful wrist), which will subsequently be the wrist used for all efficacy assessments throughout the study.

Treatment Regimen and Route of Administration: Patients will apply one patch (either a lidocaine patch 5% or a matching placebo patch) to the volar aspect of each affected wrist once every 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Are males or females 18 years of age or older
* Have confirmed diagnosis of CTS in one or both wrists. For patients with bilateral CTS, the most painful wrist will be identified as the "index" wrist, and will be the wrist used for all efficacy evaluations.
* Have clinical symptoms of pain, paresthesia, numbness and/or tingling in the distribution of the median nerve
* Have positive findings from electrodiagnostic tests using accepted criteria
* Have classification of the wrist(s) as "classic" or "probable" using the Katz Hand Diagram (Katz and Stirrat, 1990)
* Have worst daily pain intensity greater than 5 (0-10 scale) on approximately 75% of days over the previous 3 months; this criteria will be assessed at the screening visit only
* Have a normal 12-lead electrocardiogram (ECG) without any clinically significant abnormalities in heart rate, rhythm, or conduction
* Have been informed of the nature of the study and provided written informed consent

Exclusion Criteria:

* Have a positive serum pregnancy test (females of childbearing potential only)
* Have tumors or cysts in the wrist, muscle wasting in the forearm and/or hand, peripheral neuropathy, mononeuropathy multiplex, or hand arthritis
* Have had previous CTS surgery
* Have severe CTS as defined by electrodiagnostic findings
* Have had steroid injections for CTS in the previous 3 months
* Have used diuretics (except a stable dose for hypertension) or Vitamin B6 or topical treatments for CTS (e.g., ultrasound, iontophoresis, cold laser) in the past 2 weeks
* Require sleep medications
* Are using a lidocaine-containing product that cannot be discontinued during the study
* Have a known sensitivity or allergy to an amide-type local anesthetic agent para-aminobenzoic (PABA) derivatives or local anesthetics
* Have previously participated in a Lidoderm study
* Have severe renal insufficiency (creatinine clearance of <30 mL/min)
* Have moderate or greater hepatic impairment, including a history of or active hepatitis
* Have abnormal clinical laboratory test results unless deemed clinically insignificant by the investigator
* Have current or planned litigation, or who are planning to acquire or are currently receiving Worker's Compensation or Social Security benefits, or who, in the opinion of the investigator, exhibit any evidence of secondary gain (monetary or non-monetary) associated with carpal tunnel syndrome pain.
* Have a history of alcohol or substance abuse within the last 3 years
* Have received an investigational drug or product or participated in an investigational drug study within a period of 30 days or 5 half-lives prior to receiving study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2005-11; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Worst daily pain intensity score | Week 8

SECONDARY OUTCOMES:
Average daily pain intensity score | Week 8
Levine CTS Symptom Severity and Functional Status Scales | Week 8
Mean interference with daily activities | Week 8
Intensity of Various Pain Qualities | Week 8
Quality of Sleep | Week 8
Global Assessment of Treatment Satisfaction and Impression of Change | Week 8

CONTACTS AND LOCATIONS:
Overall Officials: PPD, Study Director — PPD Development, LP
Locations (1):
- PPD, Austin, Texas, United States